CLINICAL TRIAL: NCT01884818
Title: The Effect of Manipulation for Thoracic Spine Pain and Mobility, and Reliability of Used Mobility Measurements.
Brief Title: Thoracic Spine Manipulation for Patients With Thoracic Spine Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jyvaskyla (Other)
Responsible Party: Principal Investigator, Jtakatalo, Project expert, University of Jyvaskyla
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Thoracic
Record Dates: First submitted 2013-02-25; First posted 2013-06-24 (Estimated); Last update posted 2017-08-21 (Actual); Status verified 2017-08

CONDITIONS: Pain
Keywords: Thoracic spine, pain, manipulation
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Manipulation (Experimental): Subjects will receive 6 manipulation treatments within 3 weeks period. The manipulated segments are determined individually in baseline assessment.
  Interventions: Other: Manipulation vs. TNS thoracic pain
- TNS for thoracic spine (Sham Comparator): 6 TNS treatments at home for 20min in limited power of devices in three weeks period.
  Interventions: Other: Manipulation vs. TNS thoracic pain

INTERVENTIONS:
Other: Manipulation vs. TNS thoracic pain

SUMMARY:
The study includes two phases. In phase one the reliability of thoracic spine mobility measurements are studied in subjects with thoracic spine pain. In phase two the reliable measurements are used to measure the effects of thoracic spine manipulation in subjects with thoracic spine pain. The changes in pain is measured as well.

In second phase the control group receives TNS treatment six times at home as a placebo so that the power of TNS is limited to very low level. The number of treatments are controlled as well as the time of treatment. The treatment group receives six manipulation treatments within 3 week period. The effects are measured immediately after the treatment weeks, and 3 and 8 week follow-up. Moreover the one year follow-up will be performed by mail questionnaire.

DETAILED DESCRIPTION:
Outcome measures are intensity of pain (VAS, Roland-Morris questionnaire) thoracic mobility (measured with computer, tape measurements, inclinometer and manually).

ELIGIBILITY:
Inclusion Criteria:

* Thoracic spine pain,
* 18-55 years old

Exclusion Criteria:

* Inflammatory spine disease,
* previous surgery on thoracic spine area,
* osteoporosis

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2011-08; Primary Completion 2017-08-01 (Actual); Study Completion 2017-08-15 (Actual)

PRIMARY OUTCOMES:
Thoracic spine pain (Visual analogue scale) | up to 49 week follow-up

SECONDARY OUTCOMES:
Thoracic spine mobility (computer controllod spine PA measurement, tape measurements, inclinometer) | Baseline, after treatment, 3, 8, and 49 week follow-up

OTHER OUTCOMES:
Work absent | Baseline, after treatment, 3, 8 and 49 week follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Jani Takatalo, MD, Principal Investigator — University of Jyvaskyla
Locations (1):
- Fysioteekki, Oulu, Finland

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Takatalo J, Ylinen J, Pienimaki T, Hakkinen A. Intra- and inter-rater reliability of thoracic spine mobility and posture assessments in subjects with thoracic spine pain. BMC Musculoskelet Disord. 2020 Aug 10;21(1):529. doi: 10.1186/s12891-020-03551-4. PMID 32778081